CLINICAL TRIAL: NCT05208372
Title: Application of the Detection of Circulating Tumor Cell and Circulating Tumor DNA in the Diagnosis of Metastasis in Gastric Cancer
Brief Title: Detection of CTC and ctDNA in the Diagnosis of Metastasis in Gastric Cancer
Acronym: CTC_ctDNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Kai Li, Deputy Director of surgical Oncology, First Hospital of China Medical University
Other Study IDs: FirstHCMU_CTC_ctDNA
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Stomach Neoplasms; Metastasis
Keywords: Diagnosis
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparotomy group: Patients who undergo radical laparotomy for gastric cancer.
  Interventions: Diagnostic Test: CTC test; Diagnostic Test: ctDNA test
- Laparoscopy group: Patients who undergo laparoscope-assisted radical gastrectomy for gastric cancer.
  Interventions: Diagnostic Test: CTC test; Diagnostic Test: ctDNA test

INTERVENTIONS:
Diagnostic Test: CTC test — Circulating tumor cells test of ascites and blood for patients with gastric cancer.
Diagnostic Test: ctDNA test — Circulating tumor DNA test of ascites and blood for patients with gastric cancer.

SUMMARY:
To investigate the value of CTCs and ctDNA in the diagnosis of metastasis in ascites/peritoneal flushing fluid and blood; To investigate the influence of laparoscopic CO2 pneumoperitoneum establishment on peritoneal and hematogenous metastasis of advanced gastric cancer; To explore the influence of the number and type of CTCs and ctDNA on metastasis and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign informed consent.
2. Gastric cancer is determined by more than 2 pathologists.
3. Patients with Borrmann III/IV gastric cancer.

Exclusion Criteria:

1. Patients who complicate with other malignant tumors.
2. Patients who complicate with other serious heart and lung diseases.
3. Patients who receive preoperative neoadjuvant chemotherapy.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Borrmann III and Borrmann IV patients will be selected from Department of Oncology in hospitals. All patients will undergo either laparotomy or laparoscopic surgery.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Quantity of CTCs | 1 day
  To count the circulating tumor cells in ascites and blood.
Classification of CTCs | 1 day
  To classify the circulating tumor cells in ascites and blood.
Expression of ctDNA | 1 day
  To assess the expression of circulating tumor DNA in ascites and blood, including YAP1, LAMC1 and DDIT4.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Li, MD, Study Director — First Hospital of China Medical University
Locations (2):
- China (2):
  - First Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning